CLINICAL TRIAL: NCT03504566
Title: Rotation for Optimal Targeting of Albuminuria and Treatment Evaluation: A Rotation Study of Different Albuminuria Lowering Drug Classes to Study Individual Drug Response in Diabetes
Brief Title: Rotation for Optimal Targeting of Albuminuria and Treatment Evaluation (ROTATE-2)
Acronym: ROTATE-2
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Registered and published incorrectly
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Peter Rossing, Professor, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-17013487
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Diabetic Nephropathy Type 2
MeSH Terms: interventions — Linagliptin; empagliflozin; Telmisartan; glucuronyl glucosamine glycan sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): All patients recieve, in randomomized order a four way treatment schedule. Due to the nature of the study, the individual patient will serve as his/hers own comparator.
  Interventions: Drug: Linagliptin; Drug: Empagliflozin; Drug: Telmisartan; Drug: Sulodexide

INTERVENTIONS:
Drug: Linagliptin — Linagliptin
Drug: Empagliflozin — Empagliflozin
Drug: Telmisartan — Telmisartan
Drug: Sulodexide — Sulodexide

SUMMARY:
This project is an intervention study where type 2 diabetic patients will rotate through 4 different albuminuria lowering drugs with the aim to 1) quantify the individual relationship between drug exposure and albumin lowering response of different albuminuria lowering drugs in type 1 and type 2 diabetics; and 2) to investigate the effect of the same drug intervention on the glycocalyx layer in blood vessels. The overall purpose of this study is to allow for future personalized treatment of diabetics with regards to treating kidney disease more effectively than current standardized strategies.

DETAILED DESCRIPTION:
Standard treatment to patients with diabetes and persistent albuminuria nowadays are drugs inhibiting the RAAS-system as these thus assert renoprotective effects. It has been shown, that many patients do not respond to these, which means that many remain at a high renal and cardiovascular risk and highlights the need to understand the drug response variability and to find alternative albuminuria lowering treatments in order to optimize treatment for each individual.

Various drugs other than RAAS-inhibitors are available, that also decreases albuminuria. However, whether individual patients not responding to these beneficially respond to other albuminuria lowering drugs has not been prospectively investigated. Therefore a better understanding on the individual response to different albuminuria lowering drugs, of which some are developed for another indication, may help to tailor optimal therapy.

This study is designed as a randomized multicenter crossover trial with a total duration of 48 weeks and with a total of 52 patients diagnosed with type 2 diabetes, as well as elevated albuminuria (UACR between 50 mg/g and 500 mg/g).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* eGFR > 45ml/min/1.73m2
* Albumin:creatinine ratio >50mg/g and ≤500 mg/g
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Pregnant women and women of child-bearing potential who are not using reliable contraception . In addition, fertile women included in the trial must use contraceptive methods in line with the below throughout the entire trial period and until the end of relevant systemic exposure for human teratogenicity/fetal toxicity. Approved contraceptives are intrauterine devices, hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release).
* Cardiovascular disease: myocardial infarction, angina pectoris, percutaneous transluminal coronary angioplasty, coronary artery bypass grafting, stroke, heart failure (NYHA I-IV) < 6 months before inclusion
* Uncontrolled blood pressure (office BP > 160/100 mmHg)
* Active malignancy
* History of autonomic dysfunction (e.g. history of fainting or clinically significant orthostatic hypotension)
* Participation in any clinical investigation within 3 months prior to initial dosing or longer if required by local regulations, and for any other limitation of participation based on local regulations.
* Hypersensitivity to study drugs and their excipients
* Donation or loss of 400 ml or more of blood within 8 weeks prior to initial dosing
* History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during the screening.
* Any medication, surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of medications including, but not limited to any of the following:

  * Major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
  * Gastro-intestinal ulcers and/or gastrointestinal or rectal bleeding within last six months;
  * Pancreatic injury or pancreatitis within the last six months;
  * Evidence of hepatic disease as determined by any one of the following: ALT or AST values exceeding 3x ULN at inclusion visit, a history of hepatic encephalopathy, a history of esophageal varices, or a history of portocaval shunt;
  * Evidence of urinary obstruction of difficulty in voiding at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Strongest albuminuria-lowering effect. | 48 weeks
  Proportion of patients in whom the drug selected in the fifth treatment period exerts the strongest albuminuria lowering effect as compared to the other drugs used during the treatment periods.

SECONDARY OUTCOMES:
Correlation of albuminuria-lowering response. | 48 weeks
  The first secondary outcome is the degree of correlation in albuminuria-lowering responses between drugs within individual patients during the four treatment periods.
Effect on glycocalyx. | 48 weeks
  The second secondary outcome is the effect of the four drugs on the glycocalyx.

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided